CLINICAL TRIAL: NCT06847646
Title: Evaluation of Bioflex Crowns Using the Hall Technique in Primary Molars (a Randomized Controlled Clinical Trial)
Brief Title: Evaluation of Bioflex Crowns Using the Hall Technique in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yousra Ramadan, assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0931-06/2024
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: BioFlex Crowns Using Hall Technique
Keywords: BioFlex crowns; SSCs; Hall technique; TMJ function

STUDY DESIGN:
Intervention Model Description: The study was a two arm, parallel group, randomized controlled clinical trial. Allocation ratio is intended to be 1:1.
Masking Description: statistician was blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioflex crown using hall technique (Experimental): bioflex crown using the hall technique
  Interventions: Other: bioflex crown using hall technique
- stainless steel crowns using hall technique (Active Comparator): stainless steel crown using the hall technique
  Interventions: Other: stainless steel crown using hall technique

INTERVENTIONS:
Other: bioflex crown using hall technique — crowns assessment
  Arms: bioflex crown using hall technique
Other: stainless steel crown using hall technique — crown assessment
  Arms: stainless steel crowns using hall technique

SUMMARY:
The goal of this randomized controlled clinical trial is to to evaluate the clinical performance and radiographic success of BioFlex crowns versus SSCs using Hall Technique in primary dentition. The main questions it aims to answer are:

Does bioflex crowns have the same clinical performance and radiographic success of stainless steel crowns when placed using Hall Technique?

will bioflex crowns alter the occlusal vertical dimensions or affect the tempomandibular joint?

If there is a comparison group: Researchers will compare bioflex crown to stainless steel crown to see of the bioflex crowns are effective as stainless steel crowns when placed using hall technique

Participants will recieve bioflex crown and stainless steel crown according to randomization and they will be followed up immediately after treatment, after 2 weeks , after 1 months , after 3 months , after 6 months and after 12 months

DETAILED DESCRIPTION:
The study will be a double-armed randomized controlled clinical trial, with parallel design. A total of 74 pediatric patients aged 4-8 years will be selected from the Pediatric Dentistry Outpatient Clinic, Faculty of Dentistry, Alexandria University, Egypt. Participants will be allocated into 2 groups according to the type of crown used. Group I (study group) will be treated with BioFlex crowns using Hall technique, while Group II (control group) will be treated with the SSCs using Hall technique. Clinical and radiographic success of both crowns will be assessed. The function of the temporomandibular joint (TMJ) will be evaluated using the Helkimo Clinical Dysfunction Index (Di) and the AAPD questionnaire. The Occlusovertical dimension measurements will also be evaluated using the Van der Zee and Van Amerongen method. Plaque and gingival health will be recorded using plaque and gingival indices, and the satisfaction level of the child will be assessed using the Facial Image Scale (FIS), while the satisfaction level of parents will be assessed using questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Primary molar teeth with occlusal or occlusoproximal carious lesions into dentin (ICDAS codes: 3-5).

Exclusion Criteria: Teeth will be excluded if they exhibit:

* Clinical or radiographic signs of irreversible pulpitis.
* Presence of fistula or abscess.
* Spontaneous pain.
* Pulp exposure.
* Bruxism.
* Pathologic mobility (identified by gently rocking the tooth buccolingually using tweezers).

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical performance of BioFlex crowns versus SSCs using HT. | 12 months
  clinical evaluation of crown performance
  Success:
  * Satisfactory restoration/crown, no intervention required
  * No clinical signs or symptoms of pulp pathology
  Minor Failures:
  * Crown presents perforation
  * Crown loss - tooth able to be re-treated
  Major Failures:
  • Reversible or irreversible pulpitis or dental fistula/abscess, requiring pulpotomy, pulpectomy or extraction.
To evaluate the radiographic success of BioFlex crowns versus SSCs using HT. | 12 months
  radiographic evaluation using digital xrays
  • Teeth will be considered radiographically successful if they show no evidence of:
  1. Radicular radiolucency
  2. Internal or external root resorption
  3. Periodontal ligament space widening

SECONDARY OUTCOMES:
Temporomandibular joint function assessment | 6 months
  The Helkimo Clinical Dysfunction Index (modified version) assesses TMJ dysfunction based on:
  Maximum Opening:
  0 = ≥35 mm
  1. = 25-34 mm
  2. = <25 mm
  Deflection During Opening:
  0 = <2 mm
  1. = 2-5 mm
  2. = >5 mm
  Impaired TMJ Function:
  0 = no impairment
  1. = palpable click
  2. = audible click, deadlock, or luxation
  Pain in TMJ:
  0 = no pain
  1. = palpable pain
  2. = reflex pain
  Muscle Pain (Temporalis & Masseter):
  0 = no pain
  1. = palpable pain
  2. = reflex pain
  Score Classification:
  0 = no dysfunction 1-4 = mild dysfunction 5-9 = moderate dysfunction 9 = serious dysfunction
  The AAPD guidelines are used for assessing TMJ symptoms, asking about difficulty opening the mouth, pain, muscle pain in the temporalis and masseter, sounds, and jaw-related injuries. Responses are yes/no.
Changes in the occlusal vertical dimensions | 1 month
  The assessment of the OVD will be performed according to a Modified version of van der Zee and van Amerongen method The cusp tip of the left maxillary canine was marked using a pencil on the lower canine in the maximum intercuspation, and its distance to the mandibular canine cusp tip was measured using a UNC-15 probe and used as the overbite score
Dental plaque assessment | 12 months
  Criteria for scoring plaque index (Silness and Löe)
  0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pockets or the tooth and gingival margin which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and /or on the tooth and gingival margin.
gingival health assessment | 12 months
  Criteria for scoring gingival index (Löe and Silness) 0 Healthy (No gingivitis.).
  1. Mild gingivitis, Slight redness and edema, no bleeding upon probing
  2. Moderate gingivitis, moderate redness and edema, bleeding upon probing
  3. Severe gingivitis, severe redness and edema, spontaneous bleeding and ulcerations
Parental satisfaction assessment | 12 months
  • The satisfaction level of parent/legal guardian will be assessed as performed immediately post-operative, in addition to problems that the child might be facing, such as bleeding around the crown, sensitivity, and food lodgment using questionnaire Parental satisfaction will be assessed on a Likert type scale from 1 to 5 using the seven following variables: shade, size, shape, retention, durability, overall satisfaction, and child's satisfaction.
child satisfaction assessment | immediately after treatment
  • The patient's perception of the treatment will be assessed by using the Facial Image Scale (FIS) modified from the Maunuksela et al scale
  1. Very happy.
  2. Happy.
  3. Neutral.
  4. Sad.
  5. Very sad.

CONTACTS AND LOCATIONS:
Overall Officials: yousra ramadan, Ms, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry Alexandria University, Alexandria, Egypt